CLINICAL TRIAL: NCT07014215
Title: A Phase II Study Evaluating the Safety and Efficacy of Sintilimab Plus Bevacizumab and Tafolecimab in Patients With Advanced NSCLC Who Have Progressed After Anti- PD- 1/L1 Therapy
Brief Title: PD-1 Combined With Bevacizumab and PCSK-9 Inhibitor in Patients With Advanced NSCLC Who Have Progressed After Anti- PD- 1/L1 Therapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Zhihong Zhang, chief physician, Anhui Provincial Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-ethics-134
Record Dates: First submitted 2025-05-21; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-01

CONDITIONS: NSCLC (Advanced Non-small Cell Lung Cancer); Resistance to Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Drug: Sintilimab combined with bevacizumab and tafolecimab
  Interventions: Drug: Sintilimab combined with Bevacizumab and tafolecimab

INTERVENTIONS:
Drug: Sintilimab combined with Bevacizumab and tafolecimab — Patients who met the inclusion criteria were treated with sintilimab(200mg Q3W) combined with Bevacizumab(7.5mg/kg Q3W) and tafolecimab(600mg Q6W) until disease progression or intolerable adverse reactions or death(up to 24 months)

SUMMARY:
This study evaluated the sintilimab combination of bevacizumab and tafolecimab in NSCLC patients who have previously been treated with anti- PD- 1/ligand (L)1 and acquired resistance. The patients were assigned to receive sintilimab(200mg Q3W) in combination with bevacizumab(7.5mg/kg Q3W) and tafolecimab(600 mg Q6W). The primary endpoints of the study were progression- free survival (PFS) assessed by RECISTv1.1 , while secondary endpoints included objective response rate (ORR), and overall survival (OS) and safety.

ELIGIBILITY:
Inclusion Criteria:

* 1. Sign written informed consent before implementing any experimental procedures
* 2. Age ≥ 18 years old and ≤ 80 years old
* 3. Histological or cytological confirmation of locally advanced (IIIB-IIIC), metastatic or recurrent (stage IV) NSCLC (International Association for the Study of Lung Cancer and Joint Committee on Cancer Classification 9th edition TNM lung cancer staging)
* 4. Failure after previous treatment with PD - (L) 1 inhibitors (alone or in combination with another systemic therapy) (CR, PR, SD>6 months)
* 5. Previously not receiving anti angiogenic drug treatment
* 6. Confirmed by histological specimens that there are no EGFR gene sensitive mutations, ALK gene fusion mutations, ROS1 gene mutations, or RET gene mutations
* 7. According to the criteria for evaluating the efficacy of solid tumors (RECIST v1.1 version), there should be at least one measurable lesion on imaging. If the lesion located within the previous radiation field is confirmed to have progressed, it can be considered a measurable lesion
* 8. Subjects with brain metastases who are asymptomatic or have stable symptoms after local treatment are allowed to be enrolled, as long as they meet the following conditions:

  1. Measurable lesions outside the central nervous system
  2. No central nervous system symptoms or no worsening of symptoms within at least 2 weeks
  3. No need for glucocorticoid treatment, or discontinuation of glucocorticoid treatment within 7 days prior to the first dose, or stable and reduced glucocorticoid dosage to below 10mg/day of prednisone (or equivalent dose) within 7 days prior to the first dose
* 9. Subjects are allowed to receive palliative radiation therapy (including cranial radiation therapy for symptomatic brain metastases), provided that the radiation therapy is completed at least one week before enrollment and the radiation related toxicity has recovered to less than or equal to degree 1 (CTCAE 5.0, except for hair loss)
* 10. ECOG rating 0-1 points
* 11. Expected survival time>3 months
* 12. Adequate organ function, subjects must meet the following laboratory indicators:

  1. In the past 14 days without using granulocyte colony-stimulating factor, the absolute neutrophil count (ANC) is ≥ 1.5x10*9/L
  2. Platelets ≥ 100 × 10*9/L without blood transfusion in the past 14 days
  3. Hemoglobin>9g/dL without blood transfusion or use of erythropoietin in the past 14 days
  4. Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
  5. Aspartate transaminase (AST) and alanine transaminase (ALT) levels should be ≤ 2.5 × ULN (subjects with liver metastases are allowed to have ALT or AST levels ≤ 5 × ULN)
  6. Blood creatinine ≤ 1.5 × ULN and creatinine clearance rate (calculated using Cockcroft Gault formula) ≥ 60 ml/min
  7. Good coagulation function, defined as International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 times ULN
  8. Normal thyroid function is defined as thyroid stimulating hormone (TSH) within the normal range. If the baseline TSH exceeds the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can also be enrolled
  9. The myocardial enzyme spectrum is within the normal range (simple laboratory abnormalities that are deemed clinically insignificant by the researchers are also allowed to be included)
* 13. For female subjects of childbearing age, a urine or serum pregnancy test with negative results should be conducted within 3 days prior to the first administration of the study drug (Day 1 of the first cycle). If the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required. Non childbearing women are defined as those who have been postmenopausal for at least one year or have undergone surgical sterilization or hysterectomy
* 14. If there is a risk of conception, all subjects (regardless of gender) must use contraceptive measures with an annual failure rate of less than 1% throughout the entire treatment period until 120 days (or 180 days) after the last administration of the study drug

Exclusion Criteria:

* 1. Pathological diagnosis of small cell lung cancer (SCLC), including lung cancer mixed with SCLC and NSCLC
* 2. The patient has received first-line or more PD - (L) 1 inhibitor monotherapy or combination chemotherapy treatment
* 3. Received the following treatments:

  1. Received systemic anti-tumor therapy within 3 weeks prior to treatment, such as chemotherapy, targeted therapy, immunotherapy (including herbal therapy with anti-tumor indications), etc
  2. Received any investigational drug treatment within 4 weeks prior to treatment
  3. Received high doses of immunosuppressive drugs (systemic corticosteroids exceeding 10mg/day, prednisone or its equivalent) within 4 weeks prior to treatment
  4. Received attenuated live vaccine within 4 weeks prior to treatment (or planned to receive attenuated live vaccine during the study period)
  5. Has undergone major surgery (such as open cavity, thoracotomy, or Kaifu surgery) within 4 weeks before treatment, or has unhealed surgical wounds, ulcers, or fractures
* 4. There is clinically uncontrollable pleural/peritoneal effusion (subjects who do not require drainage or have no significant increase in effusion after stopping drainage for 3 days can be enrolled)
* 5. Subjects who have received chest radiation therapy greater than 30 Gy within the 6 months prior to treatment or palliative radiation therapy with a dose of 30 Gy or less within the 7 days prior to treatment (palliative radiation therapy for bone lesions or intracranial lesions is allowed)
* 6. Within 2 years prior to the first administration, there has been an active autoimmune disease requiring systemic treatment (such as the use of disease relieving drugs, corticosteroids, or immunosuppressants). Alternative therapies (such as thyroid hormone, insulin, or physiological glucocorticoids used for adrenal or pituitary insufficiency) are not considered systemic treatments
* 7. Known allogeneic organ transplantation (excluding corneal transplantation) or allogeneic hematopoietic stem cell transplantation
* 8. Individuals known to be allergic to the active ingredients or excipients of the study drug
* 9. Before starting treatment, if there has been no sufficient recovery from toxicity and/or complications caused by any intervention measures (i.e. ≤ grade 1 or baseline, excluding fatigue or hair loss)
* 10. Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive)
* 11. Untreated active hepatitis B (defined as HBsAg positive and HBV-DNA copy number detected is greater than the upper limit of normal value in the laboratory of the research center) Note: Those who meet the following criteria can also be included in the group:

  1. Before the first administration, the HBV viral load was less than 1000 copies/ml (200 IU/ml), and subjects should receive anti HBV treatment throughout the entire study drug treatment period to avoid viral reactivation
  2. For subjects with anti HBc (+), HBsAg (-), anti HBs (-), and HBV viral load (-), prophylactic anti HBV treatment is not necessary, but close monitoring of viral reactivation is necessary
* 12. Active HCV infected subjects (HCV antibody positive and HCV-RNA level above the detection limit)
* 13. Administer a live vaccine within 30 days prior to the first dose (Day 1 of the first cycle) Note: It is allowed to receive inactivated vaccine for seasonal influenza within 30 days before the first administration; But it is not allowed to receive attenuated live influenza vaccine for intranasal use
* 14. Pregnant or lactating women
* 15. There are any serious or uncontrollable systemic diseases, such as:

  1. Resting electrocardiogram shows significant and difficult to control abnormalities in rhythm, conduction, or morphology, such as complete left bundle branch block, grade II or higher heart block, ventricular arrhythmia, or atrial fibrillation
  2. Unstable angina pectoris, congestive heart failure, chronic heart failure classified as NYHA ≥ 2
  3. Myocardial infarction occurred within 6 months prior to enrollment
  4. Poor blood pressure control (systolic blood pressure>140 mmHg, diastolic blood pressure>90 mmHg)
  5. A history of non infectious pneumonia requiring corticosteroid treatment within the year prior to the first administration, or current clinical active interstitial lung disease
  6. Active pulmonary tuberculosis
  7. There are active or uncontrolled infections that require systemic treatment
  8. Presence of clinically active diverticulitis, abdominal abscess, and gastrointestinal obstruction
  9. Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis
  10. Poor control of diabetes (FBG>10mmol/L)
  11. Urine routine shows urinary protein ≥++and confirms 24-hour urinary protein quantification>1.0 g
  12. Subjects with mental disorders who are unable to cooperate with treatment
* 16. Medical history or disease evidence that may interfere with the trial results, hinder the full participation of the subjects in the study, abnormal treatment or laboratory test values, or other situations that the researchers believe are not suitable for inclusion. The researchers believe that there are other potential risks that are not suitable for participation in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
PFS | 24months
  The time from the beginning of treatment to the time when the disease progresses or the patient dies from any cause

SECONDARY OUTCOMES:
ORR | 24months
  the rate of patients with PR and CR
OS | 24months
  The time from the beginning of treatment to the time when the patient dies from any cause
AE | 24months
  Safety will be evaluated by AE

IPD SHARING:
Plan to Share IPD: Undecided